CLINICAL TRIAL: NCT03136744
Title: Reducing Sedentary Behaviour: A Novel Opportunity for Managing Comorbidity in MS?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RES0026185
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Sedentary behaviour; Co-morbidity; Intervention
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sit Less with MS (Experimental): The Sit Less with MS program is based on Social Cognitive Theory (SCT) and consists of strategies that will enable people with MS to 'sit less' by frequently interrupting sitting and 'move more' by replacing sitting with light-intensity activity during waking hours.
  Interventions: Behavioral: Sit Less with MS

INTERVENTIONS:
Behavioral: Sit Less with MS — The Sit Less with MS intervention has a total duration of 16 weeks and consists of two stages: sit less and move more stages. During the first stage (sit less), we will conduct coaching sessions with participants every week and the focus will be on interrupting their sitting time every 30 minutes. Facebook and Twitter will be also used to provide information and supplement coaching sessions. During the second stage, the focus will be on encouraging the participants to move more by replacing sitting with light intensity activities frequently throughout waking hours.

SUMMARY:
Activity recommendations for the general population and those with multiple sclerosis (MS) focus on the promotion of activity that has a moderate intensity - in other words, activity intense enough to breathe heavily and sweat. Most adults do not achieve the recommended 150 minutes of moderate-intensity activity per week. Even fewer persons with MS meet the recommendations. Those with MS often have problems with walking and fatigue, thus it is not difficult to understand that moderate intensity activity is challenging. Our study will test the feasibility of a new approach focusing on activity over the whole day - promoting light activity such as standing or walking around the house while reducing prolonged sitting (sedentary behaviour). This approach is supported by research evidence showing that too much sedentary time, especially prolonged bouts of sitting, is associated with health risk factors such as obesity and cholesterol level. Recent work with persons with MS confirms that prolonged sitting is a problem for this population and emphasises the potential importance of this approach.

This study tests the feasibility of an internet-based intervention designed to decrease sedentary behaviour and to increase upright time in people with MS.

DETAILED DESCRIPTION:
Background: The health risks of sedentary behaviour or 'sitting too much' for the general population are receiving widespread media attention, with bylines that include, "comfy chairs are killing us very softly" or "don't just sit there!" Others have suggested that sitting is the new smoking! This media attention reflects the exponential growth of research on sedentary behaviour in the last 10 years [1-4]. The investigators believe that learning more about sedentary behaviour and its health risks may be particularly relevant for those with multiple sclerosis (MS). People with MS are substantially less active than persons without MS and have co-morbidities such as walking disability and fatigue that may make achieving the 'typical' moderate to vigorous intensity exercise targets very difficult. The investigators will test a new approach to activity promotion that focuses on reducing sedentary behaviour and moving more during the day. This approach is likely to be more feasible and lead to more sustainable activity behaviour change in persons with MS. It's broad applicability - to persons with MS who move well, to those who need help to walk, and perhaps only walk at home - is a major strength of this new approach. In the end, if found to be effective, it could mean that a large majority of those with MS could receive the benefits of activity that they may be missing out on if only the usual moderate to vigorous activity programme is recommended.

Purpose: The purpose of this project is to test the feasibility of a sedentary behaviour intervention program on reducing sedentary behaviour and improving co-morbidities such as walking disability and fatigue in people with MS.

Methods: Forty persons with MS will be recruited from the community (mostly from Edmonton through our collaboration with the MS Society of Alberta) and the MS Clinic (University of Alberta Campus). The participants will be involved with the study for 24 weeks, including a 16-week intervention and an 8-week follow-up. The intervention includes two 8-week stages; 1) Sit Less Stage- Interruptions to prolonged sitting, and 2) Move More Stage- Reduction in total sitting time through replacing sitting with light physical activities.

Baseline testing will consist of demographic, anthropometric, impairment and functional testing. Subsequently, participants will be set up with an activity monitor (ActivPAL) to wear for 7 days. All outcomes, including those from the ActivPAL, will be assessed at three-time points: Baseline (Week 0), Post-intervention (Week 16), and Follow-up (Week 24). However, at mid-intervention (Week 8), data will be collected only from the ActivPAL activity monitor. A log book will be used by participants to record their wake-time and sleep-time and times when they didn't wear the monitor.

Intervention: Once baseline testing is completed, in the first week of intervention a Fitbit monitor will be attached to each participant's waist, and the participants will be asked to do the activities that they normally do every day. This information will be used to determine usual activity behaviour. Also, participants will be asked to wear the Fitbit throughout the entire 16 weeks of the intervention. A program manual will be provided to the participants to guide them throughout the 16 weeks of the intervention. In addition to the program manual, participants will receive (via email) a weekly newsletter that emphasises an aspect of behaviour change from social cognitive theory and Skype chats will be conducted as well.

Analysis: Most of the feasibility outcomes will be descriptive related to recruitment (e.g., number of participants enrolled/number of participants approached) and adherence to the intervention. Descriptive statistics (mean, SD) will be used to characterize the sample. A two-way mixed factor ANOVA will be used to determine whether there are main (time, level of disability) and/or interaction effects for two primary sedentary behaviour outcomes - the average number of sedentary interruptions, and average sedentary time per day. Effect sizes will be calculated for each of the sedentary behaviour and the co-morbidity outcomes. Where clinically meaningful change benchmarks are available, we will determine if changes achieved from the intervention were clinically significant.

ELIGIBILITY:
Inclusion Criteria

* confirmed diagnosis of MS of at least one-year duration.
* Expanded Disability Status Scale (EDSS) scores between 1 and 6.5.
* stable in terms of disease modifying drugs and rehabilitation over the previous 6 months.
* relapse free within the previous 3 months.
* physically inactive, defined as insufficiently active by Godin-Shephard Leisure-Time Physical Activity Questionnaire.
* able to walk with or without a walking aid for 10 meters.

Exclusion Criteria:

• other neurological problems besides MS or medically unstable to engage in the program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of sedentary interruptions per day | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  Change in number of sedentary breaks from baseline to post-intervention and follow-up
Average sedentary time per day | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  Change in sedentary time from baseline to post-intervention and follow-up

SECONDARY OUTCOMES:
Patient Determined Disease Steps (PDDS) | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The PDDS will be used to track patient-reported impairment level from baseline to post-intervention and follow-up
Fatigue Severity Scale (FSS) | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The FSS will be used to track patient-reported fatigue level from baseline to post-intervention and follow-up
Modified Fatigue Impact Scale | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Modified Fatigue Impact Scale will be used to track the impact of fatigue from baseline to post-intervention and follow-up
Symbol Digit Modality Test | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Symbol Digit Modality Test will be used to monitor cognitive status from baseline to post-intervention and follow-up
Hospital Anxiety and Depression Scale | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Hospital Anxiety and Depression Scale will be used to monitor level of depression from baseline to post-intervention and follow-up
Short Form McGill Pain Questionnaire | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Short Form McGill Pain Questionnaire will be used to monitor level of pain from baseline to post-intervention and follow-up
Pittsburgh Sleep Quality Questionnaire | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Pittsburgh Sleep Quality Questionnaire will be used to monitor sleep quality from baseline to post-intervention and follow-up
Godin-Shephard Leisure-Time Physical Activity Questionnaire | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Godin-Shephard Leisure-Time Physical Activity Questionnaire will be used to track self-reported physical activity level from baseline to post-intervention and follow-up
6-minute Walk Test | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The 6-minute Walk test will be used to measure endurance from baseline to post-intervention and follow-up
10-meter Walk test | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The 10-meter Walk test will be used to assess gait speed from baseline to post-intervention and follow-up
Short Physical Performance Battery | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Short Physical Performance Battery will be monitor balance, walking speed, and function from baseline to post-intervention and follow-up
Quality of Life (SF-36) Questionnaire | Baseline (week 0), post-intervention (week 16), and follow-up (week 24)
  The Quality of Life (SF-36) Questionnaire will be used to monitor patient-reported quality of life from baseline to post-intervention and follow-up

OTHER OUTCOMES:
Recruitment rate | Follow-up (Week 24)
  Number of participants enrolled out of total number approached
Proportion of participants who completed the program [Adherence] | Follow-up (week 24)
  Proportion of participants who completed the program

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Manns, PhD, Principal Investigator — University of Alberta; Robert Motl, PhD, Principal Investigator — University of Alabama at Birmingham; Saeideh Aminian, PhD, Study Director — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participants de-identified data may be shared with our co-PI, Dr. Motl, with University of Alabama at Birmingham
Supporting Information: CSR
Time Frame: Data will be available for sharing after study completion by April 30, 2019.
Access Criteria: Participants data will be de-identified prior to sharing with our co-PI, Dr. Motl with University of Alabama at Birmingham.

REFERENCES:
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Background] Healy GN, Matthews CE, Dunstan DW, Winkler EA, Owen N. Sedentary time and cardio-metabolic biomarkers in US adults: NHANES 2003-06. Eur Heart J. 2011 Mar;32(5):590-7. doi: 10.1093/eurheartj/ehq451. Epub 2011 Jan 11. PMID 21224291
- [Background] Owen N, Healy GN, Matthews CE, Dunstan DW. Too much sitting: the population health science of sedentary behavior. Exerc Sport Sci Rev. 2010 Jul;38(3):105-13. doi: 10.1097/JES.0b013e3181e373a2. PMID 20577058
- [Background] van der Ploeg HP, Chey T, Korda RJ, Banks E, Bauman A. Sitting time and all-cause mortality risk in 222 497 Australian adults. Arch Intern Med. 2012 Mar 26;172(6):494-500. doi: 10.1001/archinternmed.2011.2174. PMID 22450936
- [Derived] Mehrabani G, Aminian S, Norton S, Motl RW, Manns PJ. Preliminary efficacy of the "SitLess with MS" intervention for changing sedentary behaviour, symptoms, and physical performance in multiple sclerosis. Disabil Rehabil. 2022 Oct;44(21):6374-6381. doi: 10.1080/09638288.2021.1966520. Epub 2021 Aug 25. PMID 34433359
- [Derived] Aminian S, Motl RW, Rowley J, Manns PJ. Management of multiple sclerosis symptoms through reductions in sedentary behaviour: protocol for a feasibility study. BMJ Open. 2019 Apr 1;9(4):e026622. doi: 10.1136/bmjopen-2018-026622. PMID 30940762